CLINICAL TRIAL: NCT01555788
Title: Closed Loop Artificial Pancreas Using Intraperitoneal (IP) Insulin Via DiaPort®
Brief Title: DiaPort Closed-Loop Artificial Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8829; ID-RCB : 2011-A001212-39 (Other: Afssaps)
Record Dates: First submitted 2012-02-28; First posted 2012-03-15 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2014-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes,; diaport,; artificial pancreas,; zone mpc algorithm,; ap system,; intraperitoneal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 1 diabetic population (Experimental): The only one arm (type 1 diabetic patients treated by basal-bolus insulin and external pumps) of this study will test an artificial pancreas system that uses the intraperitoneal route to deliver insulin (through DiaPort).
  Interventions: Device: Artificial Pancreas for DiaPort system with Zone-MPC algorithm

INTERVENTIONS:
Device: Artificial Pancreas for DiaPort system with Zone-MPC algorithm — Artificial pancreas system uses the intraperitoneal route to deliver insulin (through DiaPort) in type 1 diabetic patients treated by basal-bolus insulin and external pumps.

SUMMARY:
The primary purpose of this pilot study is to test an artificial pancreas system which uses the intra-peritoneal (IP) route for insulin delivery in type 1 diabetic patients.

DETAILED DESCRIPTION:
During this study, the investigators would like to evaluate the intra-peritoneal insulin delivery as a potential breakthrough method for delivering insulin within the artificial pancreas system.

The intent is to exploit the rapid action achieved by IP insulin to compensate for meals and for management of the basal insulin needs. Patients will come for two closed-loop admissions of 24 hours. The first closed-loop will be performed using subcutaneous route, whereas the second one will be performed using the intra-peritoneale route.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be aged between 18 (inclusive) and 65 years old
* Patient must have been clinically diagnosed with Type 1 diabetes mellitus for at least one year
* Patient must have been identified as presenting an indication for the DiaPort® system, i.e. showing poor glucose control under Sc insulin delivery as shown by a sustained HbA1C level > 8% and/or high blood glucose variability including recurrent hypoglycemic events. Patient will be eligible for the study because he/she will have a DiaPort implanted.
* Patient must demonstrate proper mental status and cognition for the study
* Patient must be affiliated or beneficiary of a social medical insurance
* Patient has signed informed consent form prior to study entry

Exclusion Criteria:

* Unwilling to perform repeated glucose checks, consume standardized meals, and/or take insulin as instructed
* Evidence of cardiovascular event during the previous 6 months, non stabilized retinopathy, or clinically significant screening laboratory abnormalities
* Pregnancy, breast feeding, or intention of becoming pregnant
* Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
* Patient is actively enrolled in another clinical trial or was part of study within 30 days or whose annual study income is over 4 500€
* Persons deprived of freedom, adults protected by law or vulnerable persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent with blood glucose between 3.9 and 8.0 mmol/L (79 - 144 mg/dl) | in the post prandial period (8 first hours after meal) during the in-clinic closed-loop 24-hour study period
  Percentage of time spent with blood glucose between 3.9 and 8.0 mmol/L (79 - 144 mg/dl):
  * in the basal or late postprandial period
  * in the early postprandial period (first 4 hours). All analyses will be done by using the YSI blood glucose measurements unless otherwise noted.

SECONDARY OUTCOMES:
Mean and standard deviation blood glucose | For the early postprandial period (first 4 hours after meal) and for the non-postprandial periods (from 8 hours after meal until next meal)
  All analyses will include a comparison of the results in the Intraperitoneal versus Subcutaneous study days.
Percentage of time spent in hypoglycemia with blood glucose <3.3mmol/l (60 mg/dl) | during the 2 hospitalisations period when loop is closed (for a total of 24 hours)
  All analyses will include a comparison of the results in the Intraperitoneal versus Subcutaneous study days.
Percentage of time spent in hyperglycemia | in the early postprandial period (first 4 hours after meal) and in the basal or late postprandial period (from 8 hours after meal until next meal)
  * Percentage of time spent in hyperglycemia with blood glucose >10 mmol/l (180 mg/dl) in the early postprandial period
  * and Percentage of time spent in hyperglycemia>8mmol/l (144 mg/dl) in the basal or late postprandial period All analyses will include a comparison of the results in the Intraperitoneal versus Subcutaneous study days

CONTACTS AND LOCATIONS:
Overall Officials: Eric ER RENARD, MD, PU-PH, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France